CLINICAL TRIAL: NCT03141892
Title: FreeStyle Libre Flash Glucose Monitoring System Accuracy Study
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-VAL-17164
Record Dates: First submitted 2017-05-02; First posted 2017-05-05 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Diabetes Mellitus, Type 1 and Type 2: Subjects will wear the FreeStyle Libre Flash Glucose Monitoring System and will receive no treatment except for safety purposes.
  Interventions: Device: FreeStyle Libre Flash Glucose Monitoring System

INTERVENTIONS:
Device: FreeStyle Libre Flash Glucose Monitoring System — Blood Glucose Monitoring

SUMMARY:
This is a pivotal, non-randomized, single arm, multi-center, prospective, non-significant risk study to evaluate the FreeStyle Libre Flash Glucose Monitoring System.

DETAILED DESCRIPTION:
Up to 60 subjects will be enrolled at up to six clinical research sites in the United States. Subjects will wear two Sensors of Three unique sensor lots. Each Sensor will have a paired Reader that will be given to the subject. All Readers will be masked during the study (i.e. subjects will not be able to view glucose results obtained from the Sensor on the Reader screen).

Subjects will be asked to perform at least 8 capillary Blood Glucose (BG) tests per day using the primary Reader. Interstitial glucose readings from each Sensor will be obtained with the corresponding Readers immediately following each BG test. Subjects will follow the same BG testing schedule during in-clinic visits. Subjects will be instructed to report any problems with the device.

Subjects will make seven (7) scheduled visits to the clinical study site, including the Enrollment/Screening Visit (Visit 1). Subjects will have four (4) in-clinic visits during which intravenous blood draws and YSI reference testing will occur. Each in-clinic visit is anticipated to last approximately 10 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject must have type 1 or type 2 diabetes.
* Subject must require insulin therapy through an insulin pump and/or multiple daily insulin injections (at least 3 injections daily).
* Willing to perform a minimum of 8 finger sticks per day during the study.
* Subject must be willing to fast four individual times prior to in-clinic visits, each fast lasting a minimum of eight hours.
* Subject must be able to read and understand English.
* In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
* Subject must be available to participate in all study visits.
* Subject must be willing and able to provide written signed and dated informed consent.

Exclusion Criteria:

* Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
* Subject is pregnant, attempting to conceive or not willing and able to practice birth control during the study duration (applicable to female subjects only).
* Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. Such conditions include, but are not limited to extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, redness, infection or edema.
* Subject currently is participating in another clinical trial.
* Subject has donated blood within 112 days (3.7 months) prior to the beginning of the study activities.
* Subject is anemic.
* Subject has concomitant medical condition which, in the opinion of the investigator, could interfere with the study or present a risk to the safety or welfare of the subject or study staff. Such conditions include but are not limited to:
* History of HIV, Hepatitis B or C
* Subject has X-ray, MRI or CT appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends.
* Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with type 1 or type 2 diabetes requiring multiple daily insulin injections (MDI) or continuous subcutaneous insulin infusion (CSII).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
System Performance | Approximately 32 hours
  System performance will be characterized with respect to YSI reference venous plasma sample measurements.
System related adverse device effects and serious adverse effects | Up to 42 days
  System will be characterized by Adverse Device Effects and Serious Adverse Device Effects experienced by study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara Karinka, PhD, Study Director — Abbott Diabetes Care
Locations (4):
- United States (4):
  - William Sansum Diabetes Center, Santa Barbara, California
  - Diablo Clinical Research, Walnut Creek, California
  - Rocky Mountain Diabetes & Osteoporosis Center, Idaho Falls, Idaho
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No